CLINICAL TRIAL: NCT02120521
Title: The Predictive Values of Serum STREM and Its Correlation With MNDA Monitoring in Critically Ill Patients.
Brief Title: Serum STREM and MNDA Mointoring in ICU
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman Abd Al-maksoud Yousef, Assistant Professor, Tanta University
Other Study IDs: 1637/02/13
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Sepsis .
Keywords: Sepsis and SIRS, ICU
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sepsis group: Sixty patients are critically ill with evidence of sepsis during ICU stay (sepsis group) and sixty patients are critically ill without evidence of infectious organism (SIRS group). At admission, Patients data include clinical status; SOFA score; central venous pressure; laboratory analysis and arterial blood gas analysis are measured. Routine cultures will be obtained. The attending physician will evaluate the patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU. A serum level of sTREM-1 and MNDA will be monitored.
- SIRS group: Sixty patients are critically ill without evidence of infectious organism (SIRS group). At admission, Patients data include clinical status; SOFA score; central venous pressure; laboratory analysis and arterial blood gas analysis are measured. Routine cultures will be obtained. The attending physician will evaluate the patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU. A serum level of sTREM-1 and MNDA will be monitored.

SUMMARY:
A total of 120 patients will be included in the study. Sixty patients are critically ill with evidence of sepsis during ICU stay (sepsis group) and sixty patients are critically ill without evidence of infectious organism (SIRS group). At admission, Patients data include clinical status; SOFA score; central venous pressure; laboratory analysis and arterial blood gas analysis are measured. Routine cultures will be obtained. The attending physician will evaluate the patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU. A serum level of sTREM-1 and MNDA will be monitored.

DETAILED DESCRIPTION:
A total of 120 patients will be included in the study. Sixty patients are critically ill with evidence of sepsis during ICU stay (sepsis group) and sixty patients are critically ill without evidence of infectious organism (SIRS group). At admission, Patients data include clinical status; SOFA score; central venous pressure; laboratory analysis and arterial blood gas analysis are measured. Routine cultures will be obtained. The attending physician will evaluate the patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU. A serum level of sTREM-1 and MNDA will be monitored.

At admission, patient's age, sex, weight and height were Patients data that include the clinical status; sequential organ failure assessment (SOFA) score; temperature; heart rate; respiratory rate; blood pressure; central venous pressure; laboratory analysis (complete blood count, blood urea nitrogen, blood sugar, serum sodium, potassium, calcium, aspartate aminotransferase, alanine aminotransferase, prothrombin time, albumin and CRP) and arterial blood gas analysis were measured. Routine cultures of suspected sites, blood and urine were obtained to determine the presence of infection. We attempted to maintain the patient hemoglobin level at 10-12g/dl and central venous pressure at 8-12 cmH2o. When needed, intravascular fluid replacement, blood products and inotropic or vasopressor agents were administered. Each day the attending physician evaluated all the study patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU.

The signs of sepsis were body temperature <36C° or > 38C°, tachycardia (>90 beats/min), ventilatory frequency>20 breath/min or Pco2<32mmHg (unless the patient was mechanically ventilated), a white cell count ≥12×109 litre-1 or < 4x 109 litre-1, or >10% immature neutrophils, in addition to the presence of infection. Severe sepsis is a sepsis associated with evidence of organ dysfunction , hypoperfusion, acute alteration of mental status, elevated plasma lactate, unexplained metabolic acidosis (arterial ph<7.3), hypoxaemia, prolonged prothrombin time or decrease in platelet count >50% or ≤100×109litre1, oliguria and hypotension defined as systolic arterial pressure <90mmHg or a decrease of >40mmHg. Septic shock was defined as hypotension (<90/60mmHg) in addition to sepsis syndrome persisting despite adequate fluid resuscitation and requiring intropic support

ELIGIBILITY:
Inclusion Criteria:

* The patients staying in ICU for more than 24 hours will be included in the study.

Exclusion Criteria:

* Patients received anti-inflammatory drugs or corticosteroids before admission, patients had immunosuppressive illness, patients had chronic organ failure; patients received massive blood transfusion; patients with radiation therapy and patients with previous organ transplantation will be excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 120 critically ill patients, sixty patients are critically ill with evidence of sepsis during ICU stay (sepsis group) and sixty patients are critically ill without evidence of infectious organism (SIRS group). At admission, Patients data include clinical status; SOFA score; central venous pressure; laboratory analysis and arterial blood gas analysis are measured. Routine cultures will be obtained. The attending physician will evaluate the patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU. A serum level of sTREM-1 and MNDA will be monitored.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
dynamic changes of serum sTREM-1 and MNDA | one week
  determine the dynamic changes of serum sTREM-1 and the corresponding changes of serum MNDA and their correlation in critically ill sepsis and SIRS patients.

SECONDARY OUTCOMES:
Survival in critically ill sepsis and SIRS patients | two weeks
  determine the dynamic changes of serum sTREM-1 and the corresponding changes of serum MNDA and their correlation in critically ill sepsis and SIRS patients and survival .

CONTACTS AND LOCATIONS:
Overall Officials: Ayman A Yousef, Principal Investigator — Assistant Professor
Locations (1):
- Tanta University hospitals, Tanta, Algharbyia, Egypt